CLINICAL TRIAL: NCT00138710
Title: Short-term Effects of Aromatase Inhibition in Obese Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTC-323-150405
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Hypogonadotrophic Hypogonadism; Obesity
Keywords: obesity; Hypogonadotrophic hypogonadism; aromatase inhibition
MeSH Terms: conditions — Hypogonadism; Obesity | interventions — Letrozole

INTERVENTIONS:
Drug: Letrozole (Femara)

SUMMARY:
In this study, 50 obese men with a hormonal imbalance will be treated with letrozole or placebo for six months in order to examine the effects on the hormonal balance, and on weight loss. The study will also address the side effects and psychological effects of letrozole as compared to placebo.

DETAILED DESCRIPTION:
The aim of the study is to establish the short-term efficacy and safety of aromatase inhibition in restoring and maintaining eugonadism in hypogonadotrophic hypogonadal men. Secondary aim is to detect the short-term somatic and psychological effects.

Study design: Double blind randomized placebo-controlled trial.

Treatment: 26 weeks of either letrozole or placebo. All patients will start on 1 tablet per week, dose adjustments will be performed if serum testosterone or estradiol are outside the target range. All men will be prescribed a mildly hypocaloric diet.

Endpoints: BMI, body weight, waist circumference, body composition, exercise capacity, serum levels of several hormone markers, glucose tolerance, psychological characteristics.

All patients will be measured 6 times during the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 35 and 50
* Male sex
* Ages between 20 and 50
* Serum total testosterone under 10 nmol/l
* Serum luteinizing hormone (LH) under 9 mU/l
* Serum estradiol over 40 pmol/l

Exclusion Criteria:

* Comorbidity
* Serum prostate-specific antigen (PSA) over 4.0 U/l
* Discontinuation of smoking less than six months ago
* Medication known to affect hormonal parameters

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Body weight
Body mass index (BMI)
Waist circumference
Body composition
Exercise capacity
Serum levels of hormones
Glucose tolerance
Reported side effects
Psychological characteristics (Symptom Checklist, intelligence quotient [IQ] NPV)

SECONDARY OUTCOMES:
Lipid profile
Blood counts
Bone markers
Liver enzymes

CONTACTS AND LOCATIONS:
Overall Officials: Hans de Boer, MD PhD, Principal Investigator — Rijnstate Hospital, Arnhem, the Netherlands
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands